CLINICAL TRIAL: NCT06951308
Title: Efficacy of Carbohydrate Loading in Diabetic Type 2 Patients Undergoing CABG Surgery on CPB
Acronym: CLDM-CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Mohammad Bashar Izzat, Professor of Surgery, Damascus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PhD2-2025
Record Dates: First submitted 2025-04-18; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Heart Surgery; Ischemic Heart Disease
Keywords: Enhanced recovery program; carbohydrate loading; coronary artery bypass grafting; heart surgery; postoperative recovery
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Patients who will have carbohydrate loading 2 hours before the surgery (400 ml of 12.5 maltodextrin and 400 ml of over-the-counter fruit-based lemonade)
  Interventions: Dietary Supplement: Carbohydrate loading before surgery
- Control arm (No Intervention): Patients who will have standard fasting protocol 8 hours before surgery

INTERVENTIONS:
Dietary Supplement: Carbohydrate loading before surgery — Carbohydrate loading 2 hours before the surgery (400 ml of 12.5 maltodextrin and 400 ml of over-the-counter fruit-based lemonade)
  Arms: Intervention arm

SUMMARY:
Enhanced recovery after surgery protocols aim to optimize perioperative care and improve surgical outcomes. Preoperative carbohydrate loading has demonstrated benefits in reducing insulin resistance and improving patient outcomes. While non-diabetic patients benefit from this approach, its efficacy in diabetic type 2 patients undergoing CABG remains less understood. This study aims to address this gab by evaluating the physiological and clinical outcomes for carbohydrate loading in this specific population.

DETAILED DESCRIPTION:
A randomized controlled trial comparing diabetic type 2 patients receiving carbohydrate loading with those undergoing traditional fasting protocols. Patients will be randomized to two groups; group (a) patients will have carbohydrate loading 2 hours before the surgery (400 ml of 12.5 maltodextrin and 400 ml of over-the-counter fruit-based lemonade), while group (b) patients (control group) will have standard fasting protocol 8 hours before surgery.

Aims of the study:

1. To assess the efficacy of carbohydrate loading in reducing insulin resistance in diabetic type 2 patients undergoing CABG surgeries.
2. To monitor clinical outcomes such as infection rates, ICU stay duration, and need for inotropic and vasoactive drugs.
3. To evaluate changes in inflammatory markers including CRP levels. clinical outcome

ELIGIBILITY:
Inclusion Criteria:

All diabetic type 2 patients undergoing isolated on-pump coronary artery bypass surgery.

Exclusion Criteria:

* Missing data.
* Patients outside the study period.
* Patients undergoing other cardiac surgeries.
* Patients diagnosed with type 1 diabetes mellitus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Insulin Tolerance Test (KITT) | Preoperatively and up to 72 hours postoperatively
  Short Insulin Tolerance Test (KITT) will test changes in insulin tolerance postoperatively

SECONDARY OUTCOMES:
CRP levels | Preoperatively and up to 72 hours postoperatively
  C-Reactive Protein levels in the blood
Arterial blood gases | Preoperatively and up to 72 hours postoperatively
  Changes in arterial blood gases
Operative time | Intraoperatively, skin-to-skin
  Total operative time, skin-to-skin
CPB duration | Intraoperatively, using extracorporeal circulation
  Total time spend using cardiopulmonary bypass perfusion
Blood loss | Intraoperatively and up to 72 hours postoperatively
  Blood loss and blood product usage
Number of grafts performed | Intraoperatively, skin-to-skin
  Number of grafts performed during the operation
Use of inotrops | Intraoperatively and up to 72 hours postoperatively
  Use of inotrops to support the cardiac output
Complications | Intraoperatively and up to 72 hours postoperatively
  All perioperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad B Izzat, FRCS(CTh), Study Director — Damascus University
Locations (1):
- Damascus University Cardiac Surgery Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be uploaded on a data sharing platform
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 31, 2026, and will be available permanently
Access Criteria: IPD will be open to all through a data sharing platform

REFERENCES:
- [Background] Dock-Nascimento DB, de Aguilar-Nascimento JE, Magalhaes Faria MS, Caporossi C, Slhessarenko N, Waitzberg DL. Evaluation of the effects of a preoperative 2-hour fast with maltodextrine and glutamine on insulin resistance, acute-phase response, nitrogen balance, and serum glutathione after laparoscopic cholecystectomy: a controlled randomized trial. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1):43-52. doi: 10.1177/0148607111422719. PMID 22235107
- [Background] Vermeulen MA, Richir MC, Garretsen MK, van Schie A, Ghatei MA, Holst JJ, Heijboer AC, Uitdehaag BM, Diamant M, Eekhoff EM, van Leeuwen PA, Ligthart-Melis GC. Gastric emptying, glucose metabolism and gut hormones: evaluation of a common preoperative carbohydrate beverage. Nutrition. 2011 Sep;27(9):897-903. doi: 10.1016/j.nut.2010.10.001. Epub 2011 Jan 21. PMID 21255977
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Breuer JP, von Dossow V, von Heymann C, Griesbach M, von Schickfus M, Mackh E, Hacker C, Elgeti U, Konertz W, Wernecke KD, Spies CD. Preoperative oral carbohydrate administration to ASA III-IV patients undergoing elective cardiac surgery. Anesth Analg. 2006 Nov;103(5):1099-108. doi: 10.1213/01.ane.0000237415.18715.1d. PMID 17056939
- [Background] Amer MA, Smith MD, Herbison GP, Plank LD, McCall JL. Network meta-analysis of the effect of preoperative carbohydrate loading on recovery after elective surgery. Br J Surg. 2017 Feb;104(3):187-197. doi: 10.1002/bjs.10408. Epub 2016 Dec 21. PMID 28000931
- [Background] Sokolic J, Knezevic D, Kuharic J, Medved I, Sustic A, Zupan Z, Laskarin G, Tadin T, Sotosek Tokmadzic V. Decrease of Perforin Expressing Lymphocytes after On-Pump Coronary Artery Bypass Grafting Surgery Irrespective of Carbohydrate Preoperative Oral Feeding. Heart Surg Forum. 2019 May 22;22(3):E218-E224. doi: 10.1532/hsf.2003. PMID 31237547
- [Background] Lee B, Soh S, Shim JK, Kim HY, Lee H, Kwak YL. Evaluation of preoperative oral carbohydrate administration on insulin resistance in off-pump coronary artery bypass patients: A randomised trial. Eur J Anaesthesiol. 2017 Nov;34(11):740-747. doi: 10.1097/EJA.0000000000000637. PMID 28437263
- [Background] Rapp-Kesek D, Stridsberg M, Andersson LG, Berne C, Karlsson T. Insulin resistance after cardiopulmonary bypass in the elderly patient. Scand Cardiovasc J. 2007 Apr;41(2):102-8. doi: 10.1080/14017430601050355. PMID 17454835
- [Background] Jarvela K, Maaranen P, Sisto T. Pre-operative oral carbohydrate treatment before coronary artery bypass surgery. Acta Anaesthesiol Scand. 2008 Jul;52(6):793-7. doi: 10.1111/j.1399-6576.2008.01660.x. Epub 2008 May 12. PMID 18477073
- [Background] Feguri GR, Lima PR, Lopes AM, Roledo A, Marchese M, Trevisan M, Ahmad H, Freitas BB, Aguilar-Nascimento JE. Clinical and metabolic results of fasting abbreviation with carbohydrates in coronary artery bypass graft surgery. Rev Bras Cir Cardiovasc. 2012 Jan-Mar;27(1):7-17. doi: 10.5935/1678-9741.20120004. English, Portuguese. PMID 22729296
- [Background] Feguri GR, Lima PRL, Franco AC, Cruz FRH, Borges DC, Toledo LR, Segri NJ, Aguilar-Nascimento JE. Benefits of Fasting Abbreviation with Carbohydrates and Omega-3 Infusion During CABG: a Double-Blind Controlled Randomized Trial. Braz J Cardiovasc Surg. 2019 Mar-Apr;34(2):125-135. doi: 10.21470/1678-9741-2018-0336. PMID 30916121
- [Background] Feguri GR, de Lima PRL, de Cerqueira Borges D, Toledo LR, Batista LN, E Silva TC, Segri NJ, de Aguilar-Nascimento JE. Preoperative carbohydrate load and intraoperatively infused omega-3 polyunsaturated fatty acids positively impact nosocomial morbidity after coronary artery bypass grafting: a double-blind controlled randomized trial. Nutr J. 2017 Apr 20;16(1):24. doi: 10.1186/s12937-017-0245-6. PMID 28427403
- [Background] Egger M, Davey Smith G, Schneider M, Minder C. Bias in meta-analysis detected by a simple, graphical test. BMJ. 1997 Sep 13;315(7109):629-34. doi: 10.1136/bmj.315.7109.629. PMID 9310563
- [Background] DerSimonian R, Laird N. Meta-analysis in clinical trials. Control Clin Trials. 1986 Sep;7(3):177-88. doi: 10.1016/0197-2456(86)90046-2. PMID 3802833
- [Background] Higgins JP, Altman DG, Gotzsche PC, Juni P, Moher D, Oxman AD, Savovic J, Schulz KF, Weeks L, Sterne JA; Cochrane Bias Methods Group; Cochrane Statistical Methods Group. The Cochrane Collaboration's tool for assessing risk of bias in randomised trials. BMJ. 2011 Oct 18;343:d5928. doi: 10.1136/bmj.d5928. PMID 22008217
- [Background] Savluk OF, Kuscu MA, Guzelmeric F, Gurcu ME, Erkilinc A, Cevirme D, Ogus H, Kocak T. Do preoperative oral carbohydrates improve postoperative outcomesin patients undergoing coronary artery bypass grafts? Turk J Med Sci. 2017 Dec 19;47(6):1681-1686. doi: 10.3906/sag-1703-19. PMID 29306223
- [Background] Kotfis K, Jamiol-Milc D, Skonieczna-Zydecka K, Folwarski M, Stachowska E. The Effect of Preoperative Carbohydrate Loading on Clinical and Biochemical Outcomes after Cardiac Surgery: A Systematic Review and Meta-Analysis of Randomized Trials. Nutrients. 2020 Oct 12;12(10):3105. doi: 10.3390/nu12103105. PMID 33053694
- [Background] Tran S, Wolever TM, Errett LE, Ahn H, Mazer CD, Keith M. Preoperative carbohydrate loading in patients undergoing coronary artery bypass or spinal surgery. Anesth Analg. 2013 Aug;117(2):305-13. doi: 10.1213/ANE.0b013e318295e8d1. Epub 2013 Jun 11. PMID 23757474
- [Background] Soop M, Nygren J, Thorell A, Weidenhielm L, Lundberg M, Hammarqvist F, Ljungqvist O. Preoperative oral carbohydrate treatment attenuates endogenous glucose release 3 days after surgery. Clin Nutr. 2004 Aug;23(4):733-41. doi: 10.1016/j.clnu.2003.12.007. PMID 15297112
- [Background] Braga M, Bissolati M, Rocchetti S, Beneduce A, Pecorelli N, Di Carlo V. Oral preoperative antioxidants in pancreatic surgery: a double-blind, randomized, clinical trial. Nutrition. 2012 Feb;28(2):160-4. doi: 10.1016/j.nut.2011.05.014. Epub 2011 Sep 3. PMID 21890323
- Available data/document: Study Protocol: PhD2-2025 — https://docs.google.com/document/d/1IpRJsfgeH_tvSrji9ydietlVCuID47xq/edit?usp=sharing&ouid=106245773366942496306&rtpof=true&sd=true — Open to enyone with link